CLINICAL TRIAL: NCT04774016
Title: Iron Absorption From an Iron-fortified Follow-up Formula With and Without the Addition of a Synbiotic or Human Milk Oligosaccharides: a Stable Isotope Study in 10-14 Month-old Thai Children
Brief Title: Iron Absorption From an Iron-fortified Follow-up Formula With Added Synbiotic or Human Milk Oligosaccharides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 18.15.INF
Record Dates: First submitted 2020-12-17; First posted 2021-02-26 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Iron Absorption
MeSH Terms: interventions — Synbiotics; Health Maintenance Organizations

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Test formula C (Experimental)
  Interventions: Other: Test formula C with HMOs
- Test formula B (Experimental)
  Interventions: Other: Test formula B with synbiotic
- Test formula A (Placebo Comparator)
  Interventions: Other: Test formula A without added pre- and pro-biotic

INTERVENTIONS:
Other: Test formula A without added pre- and pro-biotic — An identical formula as test formulas fortified with 2.20 mg iron as FeSO4-58 and 0.05 mg native iron per serving (235 ml), but without added pre- or probiotic.
  Arms: Test formula A
Other: Test formula B with synbiotic — Test formula fortified with 2.20 mg iron as FeSO4-57 and 0.05 mg native iron per serving (235 ml) and added synbiotic.
  Arms: Test formula B
Other: Test formula C with HMOs — Test formula fortified with 2.20 mg iron as FeSO4-54 and 0.05 mg native iron per serving (235 ml) and added HMOs.
  Arms: Test formula C

SUMMARY:
The co-primary objectives of this study are: 1) to investigate the effect adding a synbiotic (combination of a pre-and probiotic) to iron-fortified follow-up formula (FUF) on iron bioavailability, and 2) to investigate the effect adding Human Milk Oligosaccharides (HMOs) to iron-fortified FUF on iron bioavailability in 10-14 month-old Thai children.

DETAILED DESCRIPTION:
Iron stores of healthy, full-term neonates are supposed to cover iron needs for the first 4-6 months of life. After 6 months of age, requirements for absorbed iron are high, as infants need to build body iron stores and triple their body weight before the first year of life. Iron concentrations in mature breastmilk are low (~0.3 mg/L) and cannot adequately cover the high iron requirements of children between 6 and 24 months of age. Follow-up formulas (FUF) are fortified milk-based products intended for infants above 6 months of age and young children aged 1-3 years, and are widely used as a liquid part of the weaning diet to supplement the diet of young children with macro- and micronutrients. Prebiotics and probiotics are increasingly added to foods for infants and young children due to emerging evidence on possible health benefits. We recently showed that the addition of prebiotic galacto-oligosaccharides (GOS) to an iron-containing micronutrient powder increased iron absorption in Kenyan infants. To our knowledge, the effect of the combination of pre- and probiotics (synbiotic) or human milk oligosaccharides (HMOs) on iron absorption from an iron-fortified FUF has not been investigated.

Thai children (10-14 months old) will be assigned to receive FUF fortified with isotopically labelled iron as FeSO4 1) with synbiotic, 2) HMO, and 3) without added prebiotics as a reference, in random order. Besides the iron source and synbiotic or HMO, the test FUF will be identical in terms of macro- and micronutrient composition. For the secondary objectives of this study, which will have a single-group, before-after design, each infant will receive the test FUF with added synbiotic for 25 days on gut comfort and quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained from the parents/legally acceptable representative
* Child aged 40-56 weeks (± 3 weeks)
* Child exhibits no clinical signs/symptoms of chronic disease or acute illness
* Capillary Hb ≥70 g/L
* Anticipated residence in the area for the study duration
* Z-scores for weight-for-age and weight-for-length both >-3, if the infant is severely underweight or severely malnourished.
* Singleton, full-term gestation birth (≥37 weeks)
* Birth weight ≥2.5 kg and ≤4.5 kg

Exclusion Criteria:

* Child exhibits clinical signs/symptoms of chronic infectious, metabolic, genetic illness or other disease including any condition that impacts feeding or growth
* Child received vitamin and mineral supplements in the 2 weeks prior to enrollment
* Child is exclusively breastfed
* Child received antibiotic treatments in the 4 weeks prior to enrollment
* Parents or caretakers not willing/not able to comply with the requirements of the study protocol
* Child has allergy or intolerance to cows' milk protein or lactose, or severe food allergies
* Child is participating in any other interventional clinical trial that would interfere with study outcomes

Ages: 40 Weeks to 56 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Fractional Iron Absorption (FIA) from an iron-fortified follow-up infant formula with and without the addition of a synbiotic | Measured 28 days after administration of last test formula
  FIA from test formulas will be determined based on the shift of the iron isotope ratios in whole blood.
Fractional Iron Absorption (FIA) from an iron-fortified follow-up infant formula with and without the addition of a synbiotic | Measured 14 days after administration of last test formula
  FIA from test formulas will be determined based on the shift of the iron isotope ratios in whole blood.
FIA from an iron-fortified follow-up formula with and without the addition of human oligosaccharides (HMOs) | Measured 28 days after administration of last test formula
  FIA from test formulas will be determined based on the shift of the iron isotope ratios in whole blood.
FIA from an iron-fortified follow-up formula with and without the addition of human oligosaccharides (HMOs) | Measured 14 days after administration of last test formula
  FIA from test formulas will be determined based on the shift of the iron isotope ratios in whole blood.

SECONDARY OUTCOMES:
Effects of feeding an iron-fortified FUF with added synbiotic (Formula B) for 25 days on Iron status (haemoglobin [Hb]) | At baseline and last study visit (day 40)
  Change in iron status biomarkers (Hb) from baseline until last study visit (day 40)
Effects of feeding an iron-fortified FUF with added synbiotic (Formula B) for 25 days on Iron status (plasma ferritin [PF]) | At baseline and last study visit (day 40)
  Change in iron status biomarkers (PF) from baseline until last study visit (day 40)
Effects of feeding an iron-fortified FUF with added synbiotic (Formula B) for 25 days on Iron status (soluble transferrin receptor [sTfR]) | At baseline and last study visit (day 40)
  Change in iron status biomarkers (sTfR) from baseline until last study visit (day 40)
Effects of feeding an iron-fortified FUF with added synbiotic (Formula B) for 25 days on inflammation status ((C-reactive protein [CRP]) | At baseline and last study visit (day 40)
  Change in CRP from baseline until last study visit (day 40)
Effects of feeding an iron-fortified FUF with added synbiotic (Formula B) for 25 days on inflammation status (alpha-1-acid glycoprotein [AGP])) | At baseline and last study visit (day 40)
  Change in AGP from baseline until last study visit (day 40)
Effects of feeding an iron-fortified FUF with added synbiotic (Formula B) for 25 days on gastrointestinal (GI) tolerance | At baseline and last study visit (day 40)
  Change in GI tolerance based on caregiver-reported stool frequency (number of stools per day), consistency (on a scale from watery, runny, mushy soft, formed soft, hard, and difficult-to-pass stools (yes/no) from baseline until last study visit (day 40)
Effects of feeding an iron-fortified FUF with added synbiotic (Formula B) for 25 days on gut comfort | At baseline and last study visit (day 40)
  Change in gut comfort based on Gut Comfort Questionnaire to assess overall GI burden and individual GI symptoms/GI-related behaviours from baseline until last study visit (day 40)
Effects of feeding an iron-fortified FUF with added synbiotic (Formula B) for 25 days on health-related quality of life | At baseline and last study visit (day 40)
  Change in health-related quality of life, assessed by validated Infant and Toddler Quality of Life questionnaire from baseline until last study visit (day 40)
Effect of feeding an iron-fortified FUF with added synbiotic (Formula B) for 25 days on gut microbiota composition and diversity | At baseline and last study visit (day 40)
  Change in gut microbiota composition and diversity between baseline and last study visit (day 40)
Effect of feeding an iron-fortified FUF with added synbiotic (Formula B) for 25 days on fecal pH | At baseline and last study visit (day 40)
  Change in fecal pH between baseline and last study visit (day 40)
Effect of feeding an iron-fortified FUF with added synbiotic (Formula B) for 25 days on gut inflammation | At baseline and last study visit (day 40)
  Change in gut inflammation marker (calprotectin) between baseline and last study visit (day 40)
Effect of feeding an iron-fortified FUF with added synbiotic (Formula B) for 25 days on gut integrity | At baseline and last study visit (day 40)
  Change in gut integrity marker (serum intestinal fatty acid binding protein [I-FABP]) between baseline and last study visit (day 40)

CONTACTS AND LOCATIONS:
Locations (1):
- Amphawa Hospital, Samut Sakhon, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Scheuchzer P, Sinawat S, Donze AS, Zeder C, Sabatier M, Garcia-Garcera M, Ricci C, Kamontham T, Zimmermann MB, Baumgartner J. Iron Absorption from an Iron-Fortified Follow-Up Formula with and without the Addition of a Synbiotic or a Human-Identical Milk Oligosaccharide: A Randomized Crossover Stable Isotope Study in Young Thai Children. J Nutr. 2024 Oct;154(10):2988-2998. doi: 10.1016/j.tjnut.2024.08.016. Epub 2024 Aug 22. PMID 39179207